CLINICAL TRIAL: NCT06654557
Title: Effect of Adding Glycerol to Electrolyte Beverages on Fluid Balance in Healthy Euhydrated Men and Women at Rest
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2412
Record Dates: First submitted 2024-10-18; First posted 2024-10-23 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Fluid Balance
Keywords: hydration; electrolytes; glycerol; carbohtydrate; beverage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Placebo beverage (Parts 1 and 2) (Placebo Comparator)
  Interventions: Other: Placebo beverage, kiwi-strawberry flavor (Part 1 and Part 2)
- 0% carbohydrate electrolyte solution with glycerol beverage (Part 1 only) (Experimental)
  Interventions: Other: 0% carbohydrate electrolyte solution with glycerol beverage (Part 1 only)
- 0% carbohydrate electrolyte solution without glycerol beverage (Part 1 only) (Experimental)
  Interventions: Other: 0% carbohydrate electrolyte solution without glycerol beverage (Part 1 only)
- 1% carbohydrate electrolyte solution with glycerol beverage (Parts 1 and 2) (Experimental)
  Interventions: Other: 1% carbohydrate electrolyte solution with glycerol beverage (Parts 1 and 2)
- 6% carbohydrate electrolyte solution with glycerol beverage (Parts 1 and 2) (Experimental)
  Interventions: Other: 6% carbohydrate electrolyte solution with glycerol beverage (Parts 1 and 2)
- 6% carbohydrate electrolyte solution without glycerol beverage (Part 2 only) (Experimental)
  Interventions: Other: 6% carbohydrate electrolyte solution without glycerol beverage (Part 2 only)
- 2% carbohydrate electrolyte solution without glycerol beverage (Part 2 only) (Experimental)
  Interventions: Other: 2% carbohydrate electrolyte solution without glycerol beverage (Part 2 only)

INTERVENTIONS:
Other: Placebo beverage, kiwi-strawberry flavor (Part 1 and Part 2) — 9.3 oz (276 ml) aliquots 3 times for a total of 28 oz (828 ml) over a 35 min period followed by 25 min rest until Time 0 post-dose.
  Arms: Placebo beverage (Parts 1 and 2)
Other: 0% carbohydrate electrolyte solution with glycerol beverage (Part 1 only) — 9.3 oz (276 ml) aliquots 3 times for a total of 28 oz (828 ml) over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: 0% carbohydrate electrolyte solution with glycerol beverage (Part 1 only)
Other: 0% carbohydrate electrolyte solution without glycerol beverage (Part 1 only) — 9.3 oz (276 ml) aliquots 3 times for a total of 28 oz (828 ml) over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: 0% carbohydrate electrolyte solution without glycerol beverage (Part 1 only)
Other: 1% carbohydrate electrolyte solution with glycerol beverage (Parts 1 and 2) — 9.3 oz (276 ml) aliquots 3 times for a total of 28 oz (828 ml) over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: 1% carbohydrate electrolyte solution with glycerol beverage (Parts 1 and 2)
Other: 6% carbohydrate electrolyte solution with glycerol beverage (Parts 1 and 2) — 9.3 oz (276 ml) aliquots 3 times for a total of 28 oz (828 ml) over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: 6% carbohydrate electrolyte solution with glycerol beverage (Parts 1 and 2)
Other: 6% carbohydrate electrolyte solution without glycerol beverage (Part 2 only) — 9.3 oz (276 ml) aliquots 3 times for a total of 28 oz (828 ml) over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: 6% carbohydrate electrolyte solution without glycerol beverage (Part 2 only)
Other: 2% carbohydrate electrolyte solution without glycerol beverage (Part 2 only) — 9.3 oz (276 ml) aliquots 3 times for a total of 28 oz (828 ml) over a 35 min period followed by 25 min rest until Time 0 post-dose. Beverage matched to placebo for color and flavor.
  Arms: 2% carbohydrate electrolyte solution without glycerol beverage (Part 2 only)

SUMMARY:
The results of a prior study PEP-2311 suggested there was a positive dose-response effect of glycerol and sodium on fluid balance and fluid retention. In addition, inclusion of glycerol resulted in an upward shift in the relationship between sodium concentration and fluid balance. The practical interpretation is that addition of glycerol enables a reduction in sodium concentration compared with a 0% glycerol drink.

In this follow-up study, the investigators hypothesize that 1) fluid balance will be sustained (greater than or not different from baseline) and significantly greater than placebo for 120 min after drinking the test no/low/moderate carbohydrate beverages and 2) fluid balance will not differ between the carbohydrate-electrolyte beverages, but both will be greater than placebo.

DETAILED DESCRIPTION:
This is a two-part study. Subjects will be asked to complete either Part 1 or Part 2 of this study. Subjects can participate in both parts of the study if they are interested and available to complete all trials. However, they will be asked to complete Part 1 before enrolling in Part 2 of the study. Dosing days are separated by 2-15 days.

Objective 1) To compare the effect of consumption of four no/low/moderate carbohydrate drinks with high electrolyte concentrations vs. placebo on fluid balance at rest. To enroll N=25

Objective 2) To compare the effect of consumption of two moderate carbohydrate drinks with low electrolyte concentrations vs. placebo on fluid balance at rest. To enroll N=70

ELIGIBILITY:
Inclusion Criteria:

Subject is male or female

* If female, subject is not pregnant (based on self-report)
* Subject is 18-50 years of age, inclusive Subject is at least recreationally active (engaged in light to moderate intensity, intermittent, or steady-state exercise at least 3 days per week for at least 30 min at a time)
* Subject does not smoke (or has quit for at least 6 months)
* Subject is not taking medication that may interfere with the study (e.g., diuretics)
* Subject has no health conditions that would interfere with the study, As indicated on the general health questionnaire (GHQ), e.g. cardiovascular, renal, or metabolic diseases
* Subject is not allergic to adhesives (e.g., medical tape)
* Subject is not allergic to kiwi-strawberry flavoring
* Subject is willing to avoid alcohol consumption 24 hours prior to visit(s)
* Subject is willing to fast overnight (~8-12 hours)
* Subject is willing to refrain from vigorous exercise for 24 hours (light physical activity only)
* Subject is willing to eat the exact same food the day prior to each visit to the laboratory
* Able to speak, write, and read English
* Provision of written consent to participate

Exclusion Criteria:

* Subject has participated in a clinical trial within the past 30 days
* Subject has participated in any PepsiCo trial within past 6 months
* Subject has a condition or is taking medication that the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the person at undue risk
* Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If subject is unsure if a company would be considered a competitor to Gatorade, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Fluid balance (Body Weight) | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Platform scale to the nearest 0.005 kilograms (kg)
Fluid balance (Percent (%) change in Body Mass) | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Platform scale to the nearest 0.005 kilograms (kg)

SECONDARY OUTCOMES:
Fluid retention | % change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Platform scale to the nearest 0.005 kilograms (kg), unit percent (%)
Urine mass | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Graduated cylinder on scale to the nearest 0.01 grams
Urine specific gravity | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  USG digital pen refractometer (Atago), no unit
Blood sodium | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Fingerstick sampling, unit millimoles per liter (mmol/L), iSTAT Blood Electrolyte and Chemistry Analyzer (CHEM8+ cartridge)
Blood glucose | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Fingerstick sampling, unit milligrams per deciliter (mg/dl), iSTAT Blood Electrolyte and Chemistry Analyzer (CHEM8+ cartridge)
Percent change in plasma volume | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Fingerstick sampling, calculated from hematocrit and hemoglobin concentration percent (%)
Serum glycerol concentration | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Fingerstick sampling unit millimoles per liter (mmol/L) using Sigma Aldrich glycerol assay kit
Serum osmolality | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Fingerstick sampling, unit milliosmoles per kilogram of water (mOsm/Kg H20)
Saliva osmolality | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Measured directly from the tongue using a handheld MX3 Diagnostics device, unit milliosmoles per kilogram of water (mOsm/kg H2O)
Blood pressure (systolic/diastolic) | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Automatic sphygmomanometer unit millimeters of mercury (mm/Hg)
Heart rate | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Heart rate monitor, unit beats per minute (bpm)
Subjective measure of headache | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  One item on a 100 point visual analog scale anchored from 0=No headache to 100=Severe headache
Subjective measure of lightheadedness | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  One item on a 100 point visual analog scale anchored from 0=No lightheadedness to 100=Severe lightheadedness
Subjective measures of gastrointestinal discomfort | Change each test day from pre-beverage baseline (-60 minutes) to post-beverage Time 0 minutes, 30 minutes, 60 minutes, 90 minutes,120 minutes, and 150 minutes post 3rd (last) beverage
  Eight items on a 100 point visual analog scale (stomach upset, nausea, burping, stomach bloating, abdominal discomfort, stomach fullness, vomiting, diarrhea anchored frrom 0= None to 100=Severe
Menstrual categorization | Assessed at Screening Visit
  Using Elliott-Sale chart, 2023 to categorize menstrual/hormonal contraceptive status for those who have not yet reached perimenopause/menopause. This is a decision-tree chart, not a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Baker, PhD, Principal Investigator — PepsiCo R&D Life Sciences, Sports Science
Locations (1):
- PepsiCo R&D, Gatorade Sports Science Institute, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No